CLINICAL TRIAL: NCT06761911
Title: A Real-world Study of Brentuximab Vedotin Monotherapy and Combination Regimens in the Treatment of Relapsed/Refractory Hodgkin Lymphoma
Brief Title: BV in the Treatment of Relapsed/refractory Hodgkin Lymphoma
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiuhua Sun (Other)
Responsible Party: Sponsor-Investigator, Xiuhua Sun, Head of Lymphoma and Head and Neck Oncology, Dalian Medical University
Organization: Dalian Medical University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DalianMU
Record Dates: First submitted 2024-11-12; First posted 2025-01-07 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-11

CONDITIONS: Hodgkin Lymphoma (Category)
Keywords: Brentuximab Vedotin; Hodgkin lymphoma; refractory recurrence; real world; china
MeSH Terms: conditions — Hodgkin Disease; Recurrence | interventions — Brentuximab Vedotin; sintilimab; tislelizumab; Bendamustine Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- BV monotherapy group (Active Comparator): It was initially planned that BV monotherapy would be divided into two groups: a 2-week (2W) dosing group and a 3-week (3W) dosing group. The specific dosing method was determined by the investigator, but the duration of dosing could not exceed 1 year.
  Interventions: Drug: Brentuximab Vedotin (Bv)
- BV combined treatment group (Active Comparator): For the combined treatment group, it is recommended to use drugs with low neurotoxicity, such as bendamustine and gemcitabine, and dacarbazine and etoposide can also be selected. Anti-pd-1 monoclonal antibody is recommended to be administered once every 3 weeks, and sintilimab or somatorellimab can be selected. Patients who had failed previous treatment with anti-PD-1 anti-PD-1 monoclonal antibody could also be enrolled, at the discretion of the investigator.
  Interventions: Drug: Brentuximab Vedotin (Bv); Drug: Sintilimab; Drug: Tislelizumab; Drug: Bendamustine

INTERVENTIONS:
Drug: Brentuximab Vedotin (Bv) — 1.2mg/kg/2w or 1.8mg/kg/3w
  Other Names: BV; Adcetris
Drug: Sintilimab — 200mg/3w
  Other Names: TYVYT
  Arms: BV combined treatment group
Drug: Tislelizumab — 200mg/3w
  Other Names: TEVIMBRA
  Arms: BV combined treatment group
Drug: Bendamustine — 90mg/m2/3w
  Arms: BV combined treatment group

SUMMARY:
The goal of this clinical trial is to explore the real-world Chinese relapsed/refractory patients to evaluate the efficacy and safety of BV monotherapy or combination therapy in CHL patients. The main questions it aims to answer are:

To evaluate the efficacy and toxicity of BV-containing regimen in relapsed/refractory CHL patients in China, and to provide reference for the rational and safe use of BV in clinical practice.

DETAILED DESCRIPTION:
Part I: Retrospective study The clinical data of 50 cases of relapsed/refractory CHL treated with BV in multiple centers in the past 3 years were collected. Statistical methods were used to compare the efficacy and safety between groups and subgroups.

Part II: Prospective study The study was conducted in about 20 centers in China. The preliminary plan was to select a large grade A tertiary hospital with lymphoma specialty center as a sub-center, and an investigator meeting was held to further discuss the choice of drug administration and combination therapy for patients. It was initially planned that BV monotherapy would be divided into two groups: a 2-week (2W) dosing group and a 3-week (3W) dosing group. The specific dosing method was determined by the investigator, but the duration of dosing could not exceed 1 year. For the combined treatment group, it is recommended to use drugs with low neurotoxicity, such as bendamustine and gemcitabine, and dacarbazine and etoposide can also be selected. Anti-pd-1 monoclonal antibody is recommended to be administered once every 3 weeks, and sintilimab or somatorellimab can be selected. Patients who had failed previous treatment with anti-PD-1 anti-PD-1 monoclonal antibody could also be enrolled, at the discretion of the investigator. PET-CT is recommended for efficacy evaluation, and enhanced CT can also be used for patients with poor economic conditions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically, classical hodgkin lymphoma（cHL） was diagnosed and relapsed or refractory.
* Patients were treated with BV-containing regimen at least once
* Presence of tumor (measurable or nonmeasurable).
* Signature of the form consent for participation in the study.

Exclusion Criteria:

* <18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-12-31 (Estimated); Primary Completion 2025-12-17 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Preliminary Overall Response Rate (ORR) | Up to 16 cycles (each cycle is 21 days)
  Will be calculated and a 95% confidence interval will be estimated using the Clopper-Pearson method. Assessed per Lugano 2014 Criteria at any time point while on study therapy.
Progression-free survival (PFS) | From time of study enrollment until first documentation of progressive disease or death from any cause, assessed up to 3 years
  Will be described using the Kaplan-Meier methodology. 95% confidence intervals for 1-year PFS will be calculated, with standard errors estimated using the Greenwood formula. Patients alive without disease progression will be censored at last follow-up date.

SECONDARY OUTCOMES:
Safety and tolerability of Brentuximab Vedotin | 1 year
  Adverse reactions after application of BV-containing regimen, especially hematologic toxicity

IPD SHARING:
Plan to Share IPD: No